CLINICAL TRIAL: NCT01358084
Title: NGR019: Randomized Double-blind Phase II Study of NGR-hTNF Versus Placebo as Maintenance Treatment in Patients With Advanced Malignant Pleural Mesothelioma (MPM)
Brief Title: Phase II Study of NGR-hTNF Versus Placebo as Maintenance Treatment in Patients With Advanced MPM
Acronym: NGR019
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AGC Biologics S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NGR019; 2010-023614-31 (EudraCT Number)
Record Dates: First submitted 2011-05-19; First posted 2011-05-23 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Advanced Malignant Pleural Mesothelioma
Keywords: Malignant Pleural Mesothelioma; MPM; Maintenance treatment; NGR-hTNF
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — tumor necrosis factor-alpha, CNGRC fusion protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A: NGR-hTNF + Best Supportive Care (Experimental): NGR-hTNF + Best Supportive Care
  Interventions: Drug: NGR-hTNF; Other: Best Supportive Care
- Arm B: Placebo + Best Supportive Care (Placebo Comparator): Placebo + Best Supportive Care
  Interventions: Drug: Placebo; Other: Best Supportive Care

INTERVENTIONS:
Drug: NGR-hTNF — NGR-hTNF: 0.8 mcg/m² as 60-minute intravenous infusion every week until confirmed evidence of disease progression or unacceptable toxicity occurs
  Arms: Arm A: NGR-hTNF + Best Supportive Care
Drug: Placebo — Placebo: 0.8 mcg/m² as 60-minute intravenous infusion every week until confirmed evidence of disease progression or unacceptable toxicity occurs
  Arms: Arm B: Placebo + Best Supportive Care
Other: Best Supportive Care — Where applicable and as appropriate according to Institutional clinical practice and literature guidelines. Best supportive care includes antibiotics, analgesics, antiemetics, thoracentesis, pleurodesis, blood transfusions, nutritional support, and focal external-beam radiation for control of pain, cough, dyspnea, or hemoptysis

SUMMARY:
The main objective of the trial is to document the efficacy of NGR-hTNF administered as maintenance treatment at 0.8 µg/m2 weekly in advanced malignant pleural mesothelioma

DETAILED DESCRIPTION:
First-line treatment of advanced malignant pleural mesothelioma (MPM) is based on six cycles of a pemetrexed-based chemotherapy, with a median progression-free survival (PFS) of approximately 6 months.However, the median time from completion of first-line treatment to initiation of second-line therapy is approximately 3 months. Recent experiences in non-small cell lung cancer patients have shown that a maintenance treatment given immediately after first-line treatment regimens can improve PFS and survival. Considering the toxicity profile of NGR-hTNF characterized by mild-to-moderate constitutional symptoms registered in a phase II trial in previously treated MPM patients, as well as the disease control observed in about half of the patients and maintained for more than four months and more than nine months in the triweekly and weekly cohorts, respectively, seems justified to compare in a randomized phase II trial the time-related efficacy of NGR-hTNF against placebo in advanced MPM patients who did not progress after six cycles of a standard pemetrexed-based treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Histologically or cytological confirmed malignant pleural mesothelioma of any of the following subtype: epithelial, sarcomatoid, mixed, or unknown
* Patients with non-progressive disease after six cycles of first-line, pemetrexed-based regimen administered for advanced or metastatic disease
* ECOG Performance Status 0 - 1
* Life expectancy of ≥ 12 weeks
* Adequate baseline bone marrow, hepatic and renal function, defined as follows:

  1. Neutrophils ≥ 1.5 x 109/L; platelets ≥ 100 x109/L; hemoglobin ≥ 9 g/dL
  2. Bilirubin ≤ 1.5 x ULN
  3. AST and/or ALT ≤ 2.5 x ULN in absence of liver metastasis or ≤ 5 x ULN in presence of liver metastasis
  4. Serum creatinine < 1.5 x ULN
* Measurable or non-measurable disease according to malignant pleural mesothelioma-modified RECIST criteria
* Patients may have had prior therapy providing the following conditions are met:

  * Surgery: wash-out period of 14 days
  * Radiation therapy: wash-out period of 28 days
  * Chemotherapy: wash-out period of 21 days
* Patients must give written informed consent to participate in the study

Exclusion Criteria:

* Patients must not receive any other investigational agents while on study
* Patients with myocardial infarction within the last six months, unstable angina, New York Heart Association (NYHA) grade II or greater congestive heart failure, or serious cardiac arrhythmia requiring medication
* Uncontrolled hypertension
* QTc interval (congenital or acquired) > 450 ms
* History or evidence upon physical examination of Central Nervous System disease unless adequately treated
* Patients with active or uncontrolled systemic disease/infections or with serious illness or medical conditions, which is incompatible with the protocol
* Known hypersensitivity/allergic reaction to human albumin preparations or to any of the excipients
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol
* Pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2011-03; Primary Completion 2018-12-05 (Actual); Study Completion 2018-12-05 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | every 6 weeks
  Defined as the time from the date of randomization until disease progression, or death

SECONDARY OUTCOMES:
Overall survival (OS) | every 6-12 weeks
  Defined as the time from the date of randomization until the date of death due to any cause or the last date the patient was known to be alive
Tumor response | every 6 weeks
  Assessed according to modified RECIST criteria for MPM
Safety and Toxicity according to NCI-CTCAE criteria(version 4.03) | during the study
  To evaluate safety and toxicity profile related to NGR-hTNF
Quality of life assessment by using a questionnaire according to Lung Cancer Symptom Scale (LCSS) | From date of randomization until the end of treatment, assessed every 6 weeks
  To assess changes in quality of life (QoL) in the two treatment arms.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Lambiase, MD, Study Director — AGC Biologics S.p.A.
Locations (15):
- Germany (2):
  - Zentralklinik Bad Berka GmbH, Bad Berka, Thuringia
  - Asklepios Fachkliniken München-Gauting, München-Gauting
- Italy (12):
  - Ospedale Santo Spirito, Casale Monferrato, Alessandria
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori-IRST, Meldola, Forlì-Cesena
  - Istituto Clinico Humanitas, Rozzano, Milan
  - Azienda Ospedaliera SS. Antonio e Biagio e Cesare Arrigo di Alessandria, Alessandria
  - IRCCS Azienda Ospedaliera Universitaria San Martino IST Istituto Nazionale per la Ricerca sul Cancro, Genoa
  - Asl 3 genovese, Ospedale Villa Scassi, Genova
  - IRCCS Ospedale San Raffaele, Milan
  - Istituto Oncologico Veneto, Padua
  - Azienda Ospedaliero-Universitaria di Parma, Parma
  - IRCCS Policlinico S. Matteo, Pavia
  - Azienda Unità Sanitaria locale di Ravenna, Ravenna
  - Ospedale Ca' Foncello, Treviso
- Saint Petersburg State Medical University n.a. I. P. Pavlov, Saint Petersburg, Russia